CLINICAL TRIAL: NCT06844422
Title: Adapted Guided Stereotactic Body Radiotherapy Combined with Chemotherapy and Enhancement of Novel Drug Ivonescimab for Pancreatic Cancer (ASCEND) -A Single-Arm Phase Ib/II Trial
Brief Title: Adapted Guided Stereotactic Body Radiotherapy Combined with Chemotherapy and Enhancement of Novel Drug Ivonescimab for Pancreatic Cancer (ASCEND)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Department Radiation Oncology, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-414-02
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
Keywords: Adapted Guided Stereotactic Body Radiotherapy; Chemotherapy; Ivonescimab; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: In the Phase Ib portion, a dose-escalation design using the 3 + 3 methodology will be employed over a 4-week period to establish the RP2D for Ivonescimab. The goal is to identify the optimal dose that can be safely administered to patients without excessive toxicity. Once the RP2D is determined, the trial will proceed to Phase II.
  Phase II will evaluate the efficacy of Ivonescimab at the RP2D in combination with SBRT and chemotherapy, with the primary endpoint being the median progression-free survival (mPFS) of patients with LAPC. Initially, participants will receive Ivonescimab combined with SBRT (25-50 Gy in 5 fractions) over two weeks. Following this, they will undergo up to 8-10 cycles of Ivonescimab in combination with modified FOLFIRINOX chemotherapy, which includes oxaliplatin, irinotecan, leucovorin, and fluorouracil.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic Body Radiotherapy Combined with Chemotherapy and Enhancement of Novel Drug Ivonescimab (Experimental): 1. Phase Ib (Dose Escalation):
     In this phase, patients will receive Ivonescimab in escalating doses, with the aim of determining the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and the recommended Phase II dose (RP2D). The dose-escalation process will follow a 3+3 design over a 4-week period to establish the RP2D of Ivonescimab.
  2. Phase II (Efficacy Evaluation):
  After establishing the RP2D, patients will receive Ivonescimab combined with SBRT and modified FOLFIRINOX chemotherapy.
  Interventions: Drug: Ivonescimab

INTERVENTIONS:
Drug: Ivonescimab — 1. Phase Ib (Dose Escalation):
     In this phase, patients will receive Ivonescimab in escalating doses, with the aim of determining the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and the recommended Phase II dose (RP2D). The dose-escalation process will follow a 3+3 design over a 4-week period to establish the RP2D of Ivonescimab.
  2. Phase II (Efficacy Evaluation):
  After establishing the RP2D, patients will receive Ivonescimab combined with SBRT and modified FOLFIRINOX chemotherapy.
  Other Names: Adapted Guided Stereotactic Body Radiotherapy; Chemotherapy

SUMMARY:
This study aims to evaluate the safety and efficacy of Ivonescimab, a bispecific antibody targeting PD-1 and VEGF, in combination with stereotactic body radiotherapy (SBRT) and chemotherapy for treating locally advanced pancreatic cancer (LAPC). The Phase Ib portion is a dose-escalation study to determine the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and the recommended Phase II dose (RP2D) of Ivonescimab. The Phase II portion will assess the median progression-free survival (mPFS) of patients receiving Ivonescimab with SBRT (25-50Gy/5F) and modified FOLFIRINOX chemotherapy. The study aims to provide critical insights into treatment options for LAPC and inform future therapeutic strategies.

DETAILED DESCRIPTION:
This study is a single-arm, Phase Ib/II clinical trial designed to evaluate the safety and efficacy of Ivonescimab, a bispecific antibody targeting both programmed cell death protein 1 (PD-1) and vascular endothelial growth factor (VEGF), in combination with stereotactic body radiotherapy (SBRT) and chemotherapy for locally advanced pancreatic cancer (LAPC). The trial will recruit 37 patients with LAPC, with Phase Ib focusing on determining the maximum tolerated dose (MTD), dose-limiting toxicity (DLT), and the recommended Phase II dose (RP2D) of Ivonescimab.

In the Phase Ib portion, a dose-escalation design using the 3 + 3 methodology will be employed over a 4-week period to establish the RP2D for Ivonescimab. The goal is to identify the optimal dose that can be safely administered to patients without excessive toxicity. Once the RP2D is determined, the trial will proceed to Phase II.

Phase II will evaluate the efficacy of Ivonescimab at the RP2D in combination with SBRT and chemotherapy, with the primary endpoint being the median progression-free survival (mPFS) of patients with LAPC. Initially, participants will receive Ivonescimab combined with SBRT (25-50 Gy in 5 fractions) over two weeks. Following this, they will undergo up to 8-10 cycles of Ivonescimab in combination with modified FOLFIRINOX chemotherapy, which includes oxaliplatin, irinotecan, leucovorin, and fluorouracil.

Patients will continue maintenance treatment with Ivonescimab based on individual tolerance for up to 12 months, or until intolerable toxicity or disease progression occurs. The study aims to assess both the safety and therapeutic efficacy of this novel combination treatment as a first-line approach for LAPC. Results from this Phase Ib/II study will provide critical data for the development of future treatment strategies for LAPC, potentially improving patient outcomes by targeting both the immune response and tumor vasculature.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically or cytologically confirmed unresectable LAPC, as defined by the 8th edition of the American Joint Committee on Cancer (AJCC);
2. Age between 18 and 80 years;
3. At least one measurable pancreatic cancer lesion, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
5. Life expectancy of at least 3 months;
6. Adequate hematological, renal, and hepatic function, as defined by the following criteria (within 14 days prior to enrollment): (1) Hemoglobin (Hb) ≥ 90 g/L; Absolute Neutrophil Count (ANC) ≥ 1.0 × 10^9/L; Platelet count (PLT) ≥ 75 × 10^9/L; (2) No significant organ dysfunction, with the following criteria: Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) or direct bilirubin ≤ ULN if total bilirubin > 1.5 × ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Alkaline phosphatase (ALP) ≤ 2.5 × ULN, or ≤ 2.5 × ULN for the liver fraction if ALP > 2.5 × ULN; Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance (using the MDRD formula) ≥ 40 mL/min if serum creatinine is > 1.5 × ULN; Urine protein < 2+, or if ≥ 2+ on dipstick, 24-hour urine protein must be < 2 g or the urine protein-to-creatinine ratio (UPC) must be < 2; International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN;
7. Ability to provide tissue and blood samples for translational research;
8. Ability to comprehend study details and provide written informed consent.

Exclusion Criteria:

1. History of any malignant tumors within the past 5 years, except for cured localized tumors;
2. Uncontrolled infections (e.g., active tuberculosis or hepatitis), uncontrolled systemic diseases, poorly controlled hypertension or diabetes, or severe comorbidities within the past six months, including myocardial infarction, cerebral embolism, or significant arrhythmias;
3. Previous treatment with drugs targeting other stimulatory or co-inhibitory T-cell receptors;
4. Prior radiotherapy within 2 weeks before enrollment;
5. Known allergy to Ivonescimab or its excipients;
6. Pregnancy or lactation;
7. Current or planned use of strong CYP3A4/5 or CYP1A2 inducers or strong CYP3A4/5 inhibitors;
8. Requirement for oral vitamin K antagonists for anticoagulation. Low-dose warfarin (≤ 2 mg/day) and other low-dose anticoagulants for maintaining central venous access or preventing deep vein thrombosis are permitted. Low-molecular-weight heparin is also permitted;
9. Conditions affecting oral medication administration, such as a history of gastrointestinal perforation or fistula within the past 6 months, history of intestinal obstruction, extensive bowel resection, Crohn's disease, ulcerative colitis, or chronic diarrhea.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2028-02-18 (Estimated); Study Completion 2028-02-18 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 1 years
  MTD is defined as the gradual increase in dose using 10 mg and 20 mg of ivonescimab to approach the maximum tolerated dose
Dose-Limiting Toxicity (DLT) | 1 years
  DLT is defined as unacceptable toxicities or adverse effects caused by a certain dose level of the drug, which prevent further dose escalation in participants.
Recommended Phase 2 Dose (RP2D) | 1 years
  The RP2D is the dose level of Ivonescimab recommended for use in Phase 2 clinical trials. This dose is typically chosen based on safety, tolerability, and preliminary efficacy data from Phase 1 trials.
Progression-Free Survival (PFS) | 3 years
  PFS defined as the time from the first dose of Ivonescimab to either the first radiographic evidence of disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  OS defined as the time from the first dose of Ivonescimab to the time of death from any cause.
Objective remission rate (ORR) | 3 years
  ORR defined as the proportion of subjects achieving a complete response (CR) or partial response (PR) among the total number of subjects, including an evaluation of both irradiated and non-irradiated lesions.
Disease control rate (DCR) | 3 years
  DCR defined as the proportion of subjects achieving CR, PR, or stable disease (SD) among the total number of subjects.
Duration of response (DOR) | 3 years
  DOR defined as the time from the first documented CR or PR to the first occurrence of progressive disease (PD) or death from any cause.
Local Control Rate (LCR) | 3 years
  LCR defined as the proportion of patients whose tumors have not progressed locally after receiving treatment.
Adverse Events (AEs) | 3 years
  AEs assessed according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng WC, Wang G, Mei Q. Ivonescimab Plus Chemotherapy in Patients With EGFR Variant Non-Small Cell Lung Cancer. JAMA. 2025 Jan 14;333(2):172. doi: 10.1001/jama.2024.23088. No abstract available. PMID 39661367
- [Background] Liu Z, Shan D, Han X. Ivonescimab Plus Chemotherapy in Patients With EGFR Variant Non-Small Cell Lung Cancer. JAMA. 2025 Jan 14;333(2):172-173. doi: 10.1001/jama.2024.23091. No abstract available. PMID 39661345
- [Background] Wang L, Luo Y, Ren S, Zhang Z, Xiong A, Su C, Zhou J, Yu X, Hu Y, Zhang X, Dong X, Meng S, Wu F, Hou X, Dai Y, Song W, Li B, Wang ZM, Xia Y, Zhou C. A Phase 1b Study of Ivonescimab, a Programmed Cell Death Protein-1 and Vascular Endothelial Growth Factor Bispecific Antibody, as First- or Second-Line Therapy for Advanced or Metastatic Immunotherapy-Naive NSCLC. J Thorac Oncol. 2024 Mar;19(3):465-475. doi: 10.1016/j.jtho.2023.10.014. Epub 2023 Oct 23. PMID 37879536
- [Background] Frentzas S, Austria Mislang AR, Lemech C, Nagrial A, Underhill C, Wang W, Wang ZM, Li B, Xia Y, Coward JIG. Phase 1a dose escalation study of ivonescimab (AK112/SMT112), an anti-PD-1/VEGF-A bispecific antibody, in patients with advanced solid tumors. J Immunother Cancer. 2024 Apr 19;12(4):e008037. doi: 10.1136/jitc-2023-008037. PMID 38642937
- [Background] Dhillon S. Ivonescimab: First Approval. Drugs. 2024 Sep;84(9):1135-1142. doi: 10.1007/s40265-024-02073-w. Epub 2024 Jul 29. PMID 39073550
- [Background] HARMONi-A Study Investigators; Fang W, Zhao Y, Luo Y, Yang R, Huang Y, He Z, Zhao H, Li M, Li K, Song Q, Du X, Sun Y, Li W, Xu F, Wang Z, Yang K, Fan Y, Liu B, Zhao H, Hu Y, Jia L, Xu S, Yi T, Lv D, Lan H, Li M, Liang W, Wang Y, Yang H, Jia Y, Chen Y, Lu J, Feng J, Liu C, Zhou M, Zhou J, Liu X, Zhou N, He M, Dong X, Chen H, Chen Y, Su H, Li X, Zhang Z, Yang L, Cheng Y, Chen L, Hou X, Zhang Y, Guo J, Wang Z, Lu H, Wu D, Feng W, Li W, Huang J, Wang Y, Song X, Peng J, Liu L, Guo Y, Li W, Lu D, Hu M, Wang ZM, Li B, Xia M, Zhang L. Ivonescimab Plus Chemotherapy in Non-Small Cell Lung Cancer With EGFR Variant: A Randomized Clinical Trial. JAMA. 2024 Aug 20;332(7):561-570. doi: 10.1001/jama.2024.10613. PMID 38820549